CLINICAL TRIAL: NCT01415232
Title: The Use of Ultrasound With the Epidural Depth Equation (EQ-US) to Estimate Epidural Depth (Est-D) in Morbidly Obese Parturients (BMI>40Kg/m2) Will Have a High Correlation With Actual Epidural Needle Depth (ND)
Brief Title: A Novel Way to Estimate Epidural Depth in Morbidly Obese Parturient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manuel C. Vallejo (Other)
Responsible Party: Sponsor-Investigator, Manuel C. Vallejo, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PRO10070214
Record Dates: First submitted 2011-08-09; First posted 2011-08-11 (Estimated); Results first posted 2013-05-03 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-09

CONDITIONS: Obesity
Keywords: Obesity; Ultrasound
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ultrasound measurement (Experimental): Ultrasound using the Sonosite S-Nerve® US system (SonoSite, Bothell,WA) to measure depth to epidural space in morbidly obese parturients.
  Interventions: Device: Sonosite S-Nerve® US system (SonoSite, Bothell,WA)

INTERVENTIONS:
Device: Sonosite S-Nerve® US system (SonoSite, Bothell,WA) — Ultrasound to measure depth to the epidural space in morbidly obese parturients
  Other Names: Ultrasound machine; Sonosite

SUMMARY:
The purpose of this study is to determine the correlation between actual epidural needle depth (ND) and the use of ultrasound with an epidural depth equation (EQ-US) to estimate epidural depth (Est-D) in morbidly obese parturients. It is well documented that in women with a BMI greater than 40 kg/m2 successful epidural placement is more difficult. To the best of our knowledge the use of an epidural depth equation, which was developed in an earlier study using height and weight, with ultrasound visualization will improve identification of the epidural space.

DETAILED DESCRIPTION:
The investigators plan to enroll women who are morbidly obese (BMI > 40 kg/m2) and request epidural analgesia for labor. After written informed consent, 160 patients will have the use of the epidural depth equation with ultrasound (EQ-US) to estimate epidural depth (Est-D). US visualization of the epidural space will be completed by the principle investigator who has had extensive training in epidural US visualization. The EQ-US depth will be recorded. After US use, another provider who is listed as an investigator will place the epidural catheter without prior knowledge of the estimated epidural depth with the use of the equation and US. The actual needle depth to the epidural space (ND) will be recorded.

Data collected from the patient's medical record will include demographic data (age, height, weight) gravidity, parity, and cervical dilation. Measured variables will include the estimated epidural depth (Est-D) as measured by the epidural depth equation with the use of ultrasound (EQ-US), and actual epidural needle depth (ND). The investigators believe that the use of ultrasound with the epidural depth equation (EQ-US) to estimate epidural depth (Est-D) in morbidly obese parturients will have a high correlation with actual epidural needle depth (ND).

ELIGIBILITY:
Inclusion Criteria:

All women of childbearing age (including children aged 14 years and above) with a BMI > 40kg/m2 who request epidural analgesia at Magee-Womens Hospital will be eligible to participate in the study. Men will not be included since they can not become pregnant. All patients will be recruited at Magee-Womens Hospital.

Exclusion Criteria:

Patients with severe preeclampsia will be excluded from the study, as these patients may have significant edema which could alter ultrasound and/or epidural needle depth measurement. Patients with a history of back surgery, significant scoliosis, and/or lumbar pathology (i.e. Ankylosing Spondylitis) will be excluded from the study because these conditions could complicate ultrasound visualization and/or epidural needle placement.

Ages: 14 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 160 (Actual)
Dates: Start 2010-08; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manuel C. Vallejo, M.D., Principal Investigator — University of Pittsburgh
Locations (1):
- Magee-Womens Hospital, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From August 2010 to June 2011, a total of 160 parturients from Magee-Womens Hospital of UPMC.
Period: Overall Study
Arm/Group | Ultrasound Measurement
Started | 160
Completed | 160
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ultrasound Measurement
Number analyzed (Participants) | 160
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 160
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.9 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 160
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 160

OUTCOME MEASURES:

1. Primary Outcome: Correlation Between Actual Epidural Needle Depth (ND) and Estimated Epidural Depth (Est-D)
Description: Measured using the Pearson correlation coefficient between actual epidural needle depth (ND) and epidural depth as estimated by the epidural depth equation (EQ-US) followed by ultrasound (longitudinal and transverse planes) measurement.
Time Frame: at the time of labor epidural catheter insertion (an average of 5 minutes for ultrasound visualization)
Population: per protocol
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Groups:
- Ultrasound Measurement: Ultrasound using the Sonosite S-Nerve® US system (SonoSite, Bothell,WA) to measure depth from the skin to the epidural space in morbidly obese parturients
Arm/Group | Ultrasound Measurement
Number analyzed (Participants) | 160
correlation coefficient
  Ultrasound Longitudinal Plane | 0.905 [0.873 to 0.929]
  Ultrasound Transverse Plane | 0.899 [0.865 to 0.925]
Statistical Analysis 1: Comparison: Ultrasound Measurement; Pearson's correlation coefficient was calculated for epidural distance measurements which included actual clinical epidural needle depth (ND) and the epidural depth equation (EDE), ND and prior EDE + US midline longitudinal plane view, ND and prior EDE + US transverse plane view; Test type: Non-Inferiority or Equivalence — Balki et al found a Pearson's correlation coefficient between the UD and ND depth of 0.85 (95% CI 0.75-0.91). We believe EDE + US would result in a correlation coefficient of approximately 0.91. To keep the lower bound estimate within 0.04 of a correlation of 0.91, and to maintain a 95% confidence level, 140 patients would need to be sampled. To allow for patients who may not complete the study, 160 patients were enrolled; p < 0.05, longitudinal correlation coefficient; correlation coefficient = 0.91, 95% CI 2-sided [0.87 to 0.93]
Statistical Analysis 2: Comparison: Ultrasound Measurement; Transverse plane correlation coefficient; Test type: Non-Inferiority or Equivalence — correlation coefficient; p > 0.85, transverse plane correlation coefficient; transverse plane correlation coefficient = 0.90, 95% CI 2-sided [0.87 to 0.93]
Statistical Analysis 3: Comparison: Ultrasound Measurement; Clinical epidural needle depth; Test type: Superiority or Other; p > 0.05, t-test, 2 sided; Mean Difference (Final Values) = 6.64, 95% CI 2-sided [6.5 to 6.8], Standard Deviation 1.0
Statistical Analysis 4: Comparison: Ultrasound Measurement; Estimated epidural depth equation depth (cm); Test type: Superiority or Other; p > 0.05, Formula calculation; Formula calculation = 6.54, 95% CI 2-sided [6.44 to 6.65], Standard Deviation 0.68 — Estimated epidural depth equation depth (cm)

ADVERSE EVENTS:
Arm/Group | Ultrasound Measurement
Serious Adverse Events (participants affected / at risk) | 0/160
Other Adverse Events (participants affected / at risk) | 0/160

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No